CLINICAL TRIAL: NCT05977868
Title: Comparing Oral Versus Parenteral Antimicrobial Therapy (COPAT) Trial
Brief Title: Comparing Oral Versus Parenteral Antimicrobial Therapy
Acronym: COPAT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: DSMB recommendation based on safety benefit in Experimental (oral) arm
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Joy J. Juskowich, MD, Assistant Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2304754420
Record Dates: First submitted 2023-07-14; First posted 2023-08-07 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Endovascular Infection; Bone and Joint Infection; Skin and Soft Tissue Infection; Pulmonary Infection; Gastrointestinal Infection; Genitourinary Infection
Keywords: COpAT; Oral antimicrobial therapy; OPAT; Parenteral antimicrobial therapy; Intravenous antimicrobial therapy; Implementation science
MeSH Terms: conditions — Soft Tissue Infections | interventions — Amoxicillin; Amoxicillin-Potassium Clavulanate Combination; Cefadroxil; Cefpodoxime; Cephalexin; Ciprofloxacin; delafloxacin; Doxycycline; Levofloxacin; Linezolid; Metronidazole; Moxifloxacin; Rifampin; Trimethoprim, Sulfamethoxazole Drug Combination; Ampicillin; sultamicillin; Cefazolin; Cefepime; Ceftaroline; Ceftazidime; avibactam, ceftazidime drug combination; dalbavancin; Daptomycin; Ertapenem; Meropenem; oritavancin; Oxacillin; Penicillins; Piperacillin, Tazobactam Drug Combination; Tigecycline; Vancomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The primary outcome of cure at 3 months will be adjudicated by a 2 ID faculty blinded to study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental) (Experimental): COpAT (oral antimicrobial therapy) on hospital discharge
  Interventions: Drug: Amoxicillin, amoxicillin-clavulanate, cefadroxil, cefpodoxime, cefalexin, ciprofloxacin, delafloxacin, doxycycline, levofloxacin, linezolid
- Group 2 (Control) (Active Comparator): Standard of care (IV antimicrobial therapy) on hospital discharge
  Interventions: Drug: Ampicillin, ampicillin-sulbactam, cefazolin, cefepime, ceftaroline, ceftazidime, ceftazidime-avibactam, dalbavancin, daptomycin, ertapenem

INTERVENTIONS:
Drug: Amoxicillin, amoxicillin-clavulanate, cefadroxil, cefpodoxime, cefalexin, ciprofloxacin, delafloxacin, doxycycline, levofloxacin, linezolid — COpAT (oral antimicrobial therapy) on hospital discharge
  Other Names: metronidazole, moxifloxacin, rifampin, trimethoprim-sulfamethoxazole
  Arms: Group 1 (Experimental)
Drug: Ampicillin, ampicillin-sulbactam, cefazolin, cefepime, ceftaroline, ceftazidime, ceftazidime-avibactam, dalbavancin, daptomycin, ertapenem — Standard of care (IV antimicrobial therapy) on hospital discharge
  Other Names: meropenem, oritavancin, oxacillin, penicillin, piperacillin-tazobactam, tigecycline, vancomycin
  Arms: Group 2 (Control)

SUMMARY:
This is an investigator initiated multisite pragmatic randomized controlled trial designed to demonstrate equivalent effectiveness with improved safety of early transition from intravenous (IV) antimicrobial therapy to complex outpatient oral antimicrobial therapy (COpAT) across various infectious diseases (endovascular, bone and joint, skin and soft tissue, pulmonary, gastrointestinal, and genitourinary infections).

All patients referred for outpatient parenteral antimicrobial therapy (OPAT) will be evaluated by the research team with respect to inclusion/exclusion criteria. If determined eligible for enrollment, patients will be approached by a study investigator who will present the COPAT Trial. Once informed consent is obtained, patients will be randomized 2:1 using computer software into experimental or control (standard of care) group, respectively: Experimental: COpAT only on hospital discharge; Control: Conventional OPAT, OPAT transitioned to COpAT later in outpatient setting, or long-acting parenteral lipoglycopeptides. Both groups will be followed by an ID physician on the research team with in-person or telemedicine ID Clinic standard of care visits at 2, 6, and 12 weeks after hospital discharge. At the 6-week ID Clinic follow-up, patients will be asked to complete a patient satisfaction survey. The following 2 primary outcomes will be assessed: cure at 3 months using clinical (resolution of infection) and laboratory (improvement in inflammatory markers) parameters and adverse events related to antimicrobial therapy/vascular access complication or readmission at 3 months. The following secondary outcome will be assessed: patient satisfaction at 6 weeks. The experimental group is being compared to standard of care in current clinical practice.

As this is a pragmatic clinical trial, patients will not undergo additional invasive testing or procedures.

ELIGIBILITY:
Inclusion (must meet all of the following):

* English speaking
* The patient is hospitalized at J.W. Ruby Memorial Hospital, United Hospital Center, Berkeley Medical Center, Wheeling Hospital, or Camden Clark Medical Center
* The patient has been diagnosed with ≥ 1 of the following: endovascular, bone and joint, skin and soft tissue, pulmonary, gastrointestinal, or genitourinary infection
* The patient is being transitioned to 2-8 weeks of IV antibacterial therapy on hospital discharge
* The patient has capacity to participate in routine OPAT/COpAT follow-up (telephone check-ins, laboratory monitoring, and in-person or telemedicine ID Clinic follow-up)

Exclusion (may not meet any of the following):

* The patient is not appropriate for OPAT (active injection drug use, lack of infusion resources, and/or unstable outpatient environment)
* The patient is not appropriate for COpAT (unable to receive PO medication or lack of an effective PO antimicrobial option based on susceptibility testing)
* The patient is unable to give informed consent
* The patient is a prisoner, pregnant, and/or mentally handicapped
* The patient is determined unsafe for enrollment at the primary team's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joy J. Juskowich, MD, Principal Investigator — West Virginia University; Arif R. Sarwari, MD, MSc, MBA, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iversen K, Ihlemann N, Gill SU, Madsen T, Elming H, Jensen KT, Bruun NE, Hofsten DE, Fursted K, Christensen JJ, Schultz M, Klein CF, Fosboll EL, Rosenvinge F, Schonheyder HC, Kober L, Torp-Pedersen C, Helweg-Larsen J, Tonder N, Moser C, Bundgaard H. Partial Oral versus Intravenous Antibiotic Treatment of Endocarditis. N Engl J Med. 2019 Jan 31;380(5):415-424. doi: 10.1056/NEJMoa1808312. Epub 2018 Aug 28. PMID 30152252
- [Background] Li HK, Rombach I, Zambellas R, Walker AS, McNally MA, Atkins BL, Lipsky BA, Hughes HC, Bose D, Kumin M, Scarborough C, Matthews PC, Brent AJ, Lomas J, Gundle R, Rogers M, Taylor A, Angus B, Byren I, Berendt AR, Warren S, Fitzgerald FE, Mack DJF, Hopkins S, Folb J, Reynolds HE, Moore E, Marshall J, Jenkins N, Moran CE, Woodhouse AF, Stafford S, Seaton RA, Vallance C, Hemsley CJ, Bisnauthsing K, Sandoe JAT, Aggarwal I, Ellis SC, Bunn DJ, Sutherland RK, Barlow G, Cooper C, Geue C, McMeekin N, Briggs AH, Sendi P, Khatamzas E, Wangrangsimakul T, Wong THN, Barrett LK, Alvand A, Old CF, Bostock J, Paul J, Cooke G, Thwaites GE, Bejon P, Scarborough M; OVIVA Trial Collaborators. Oral versus Intravenous Antibiotics for Bone and Joint Infection. N Engl J Med. 2019 Jan 31;380(5):425-436. doi: 10.1056/NEJMoa1710926. PMID 30699315
- [Background] Pries-Heje MM, Wiingaard C, Ihlemann N, Gill SU, Bruun NE, Elming H, Povlsen JA, Madsen T, Jensen KT, Fursted K, Schultz M, Ostergaard L, Christensen JJ, Christiansen U, Rosenvinge F, Helweg-Larsen J, Fosbol EL, Kober L, Torp-Pedersen C, Tonder N, Moser C, Iversen K, Bundgaard H. Five-Year Outcomes of the Partial Oral Treatment of Endocarditis (POET) Trial. N Engl J Med. 2022 Feb 10;386(6):601-602. doi: 10.1056/NEJMc2114046. No abstract available. PMID 35139280
- [Background] Staples JA, Ho M, Ferris D, Hayek J, Liu G, Tran KC, Sutherland JM. Outpatient Versus Inpatient Intravenous Antimicrobial Therapy: A Population-Based Observational Cohort Study of Adverse Events and Costs. Clin Infect Dis. 2022 Nov 30;75(11):1921-1929. doi: 10.1093/cid/ciac298. PMID 35439822
- [Background] Rivera CG, Mehta M, Ryan KL, Stevens RW, Tucker KJ, Mahoney MV. Role of infectious diseases pharmacists in outpatient intravenous and complex oral antimicrobial therapy: Society of Infectious Diseases Pharmacists insights. J Am Coll Clin Pharm. 2021;4:1161-1169. doi: 10.1002/jac5.1473
- [Background] Juskowich JJ, Ward A, Spigelmyer AE, Howard CA, Slain D, Guilfoose JA, Edmond MB, Sarwari AR. Complex Outpatient Oral Antimicrobial Therapy (COpAT) Program at a Rural Academic Medical Center: Evaluation of First 100 Patients. Open Forum Infect Dis. 2022; 9(2): S418-S419. doi: 10.1093/ofid/ofac492.843
- [Background] Freling S, Wald-Dickler N, Banerjee J, Canamar CP, Tangpraphaphorn S, Bruce D, Davar K, Dominguez F, Norwitz D, Krishnamurthi G, Fung L, Guanzon A, Minejima E, Spellberg M, Spellberg C, Baden R, Holtom P, Spellberg B. Real-World Application of Oral Therapy for Infective Endocarditis: A Multicenter, Retrospective, Cohort Study. Clin Infect Dis. 2023 Sep 11;77(5):672-679. doi: 10.1093/cid/ciad119. PMID 36881940

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 (Experimental) | Group 2 (Control)
Started | 64 | 30
Completed (A total of 94 patients were enrolled, but four withdrew early prior to hospital discharge: two preferred oral antibiotics, one preferred IV antibiotics, and one transitioned to comfort care (mortality).) | 62 | 28
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Transitioned to comfort care | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Experimental) | Group 2 (Control) | Total
Number analyzed (Participants) | 62 | 28 | 90
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57.5 [49 to 69] | 61.5 [51.5 to 70] | 60 [50 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 8 | 33
  Male | 37 | 20 | 57
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 62 | 28 | 90
Length of Hospital Stay [Median (Inter-Quartile Range); unit: days] | 8 [6 to 11] | 10 [7 to 11] | 9 [6 to 11]
Comorbidities [Number; unit: participants]
  Obesity | 39 | 17 | 56
  Diabetes | 33 | 11 | 44
  Cardiac | 18 | 13 | 31
  Pulmonary | 10 | 5 | 15
  Renal | 6 | 0 | 6
Infection Type [Count of Participants; unit: Participants]
  Endovascular | 8 | 5 | 13
  Bone and Joint | 46 | 20 | 66
  Other | 8 | 3 | 11
Bacteremia [Count of Participants; unit: Participants] | 30 | 13 | 43
Surgery/Drainage [Count of Participants; unit: Participants] | 55 | 19 | 74
Organism Isolated [Number; unit: participants]
  Staphylococcus aureus | 38 | 17 | 55
  MRSA | 15 | 3 | 18
  MSSA | 23 | 14 | 37
  Streptococcus species | 13 | 7 | 20
  Enterobacterales | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Cure/Control at 3 Months
Description: Number of patients with cure/control using clinical (resolution of infection - e.g., wound healed) and laboratory (improvement in inflammatory markers - e.g., CRP normalization) parameters as adjudicated by 2 ID faculty blinded to study arm
Time Frame: 3 months after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Experimental) | Group 2 (Control)
Number analyzed (Participants) | 62 | 28
Participants | 61 | 28

2. Primary Outcome: Adverse Events Related to Antimicrobial Therapy
Description: Number of participants with adverse events requiring intervention related to antimicrobial therapy (e.g., thrombocytopenia)
Time Frame: Up to 3 months after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Experimental) | Group 2 (Control)
Number analyzed (Participants) | 62 | 28
Participants | 4 | 4

3. Primary Outcome: Adverse Events Related to Vascular Access
Description: Number of participants with adverse events requiring intervention related to vascular access complication (e.g., deep venous thrombosis)
Time Frame: Up to 3 months after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Experimental) | Group 2 (Control)
Number analyzed (Participants) | 62 | 28
Participants | 0 | 7

4. Primary Outcome: Overall Readmission
Description: Number of participants readmitted for any reason up to 3 months after discharge from the hospital
Time Frame: Up to 3 months after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Experimental) | Group 2 (Control)
Number analyzed (Participants) | 62 | 28
Participants | 17 | 7

5. Secondary Outcome: Number of Participants Reporting 'Satisfied' or 'Very Satisfied' on Patient Satisfaction Survey
Description: Patient satisfaction using the COPAT Trial Patient Satisfaction Survey at 6 Weeks, which is a short questionnaire (with the overall satisfaction question incorporating a Likert scale 1= Very Dissatisfied, 5= Very Satisfied) designed to assess overall patient satisfaction. Overall satisfaction totaled from participants answering 4= Satisfied and 5= Very Satisfied.
Time Frame: 6 weeks after hospital discharge
Population: Four withdrew early prior to hospital discharge: 3 chose not to participate, and one transitioned to comfort care (mortality).
Measure: Number; unit: participants
Arm/Group | Group 1 (Experimental) | Group 2 (Control)
Number analyzed (Participants) | 61 | 28
participants | 60 | 27

6. Secondary Outcome: Number of Participants Who Answered 'Yes' to the Survey Question "Would You Have Preferred to be in the Other Study Arm? (Yes or No)"
Description: The number of participants who expressed a preference to be in the other study arm (i.e., answers 'Yes' to the survey question "Would you have preferred to be in the other study arm? Yes or No").
Time Frame: 6 weeks after hospital discharge
Population: Four withdrew early prior to hospital discharge: three chose not to participate, and one transitioned to comfort care (mortality).
Measure: Number; unit: participants
Arm/Group | Group 1 (Experimental) | Group 2 (Control)
Number analyzed (Participants) | 61 | 28
participants | 1 | 21

ADVERSE EVENTS:
Time Frame: Until study completion, for a duration of up to three months after hospital discharge
Groups:
- Experimental: Discharged with oral antibiotics
- Control: Discharged with IV antibiotics
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 1/64 | 0/30
Serious Adverse Events (participants affected / at risk) | 18/64 | 7/30
Other Adverse Events (participants affected / at risk) | 4/64 | 8/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=64) | Control (N=30)
Readmission (General disorders) | 7 (7) | 2 (2)
Readmission (Surgical and medical procedures) | 6 (7) | 1 (1)
Readmission (Infections and infestations) | 3 (3) | 1 (1)
Readmission (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Readmission (Cardiac disorders) | 1 (1) | 2 (3)
Readmission (Vascular disorders) | 0 (0) | 1 (1)
Mortality (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=64) | Control (N=30)
Antibiotic Side Effect (General disorders) | 3 (3) | 2 (2)
Antibiotic Side Effect (Infections and infestations) | 1 (1) | 1 (1)
Antibiotic Side Effect (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Line Related Adverse Event (Vascular disorders) | 0 (0) | 7 (8)

LIMITATIONS AND CAVEATS:
Our trial was unblinded for pragmatic reasons. Assessment of clinical cure/control by 2 ID physicians blinded to study arm minimized potential bias. More patients in Experimental group had a procedure for source control. At least two ID physicians select oral regimens to optimize safety. Patients with active SUD/IDU were excluded. All patients were followed through OPAT and COpAT programs. Study results may not be generalizable to institutions/practices without these programs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT05977868/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT05977868/ICF_001.pdf